CLINICAL TRIAL: NCT03176628
Title: Randomized, Double-blind, Placebo-controlled, Stepwise Study of the Pharmacokinetics, Pharmacodynamics & Safety of Escalating Doses of Basis (Nicotinamide Riboside and Pterostilbene) in Patients With Acute Kidney Injury (AKI)
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of Basis in Acute Kidney Injury Study
Acronym: BAKIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Elysium Health (Industry)
Responsible Party: Principal Investigator, Eugene Rhee, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2017P000908
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Acute Kidney Injury
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Acute Kidney Injury | interventions — Radial Basis Function Networks; nicotinamide-beta-riboside; Pterocarpus marsupium

STUDY DESIGN:
Intervention Model Description: Randomized 5 subjects in active arm (Basis) : 1 subject in control (placebo)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo capsules are identical in appearance to active agent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basis (Experimental): Nicotinamide riboside (NR) and pterostilbene oral capsules 250mg/50mg (Step 1) twice daily for 2 days. If the study progresses to Steps 2, 3, and 4, then 2x, 3x, and 4x the doses in Step 1 will be administered.
  Interventions: Dietary Supplement: Basis
- Placebo (Placebo Comparator): Capsules identical in appearance and number to the agent used in Steps 1-4.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Basis — NR is a form of vitamin B3; Pterostilbene is a natural dietary compound and the primary antioxidant component of blueberries
  Other Names: nicotinamide riboside (NR) and pterostilbene
  Arms: Basis
Dietary Supplement: Placebo — Placebo capsule(s)
  Arms: Placebo

SUMMARY:
This study will determine the pharmacokinetics, pharmacodynamics and safety of escalating doses of Basis following twice daily oral administration in patients with acute kidney injury (AKI). Basis is a commercially available nutritional supplement consisting of nicotinamide riboside (NR) and pterostilbene that acts to increase sirtuin activity.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is common, growing in incidence, and associated with significant morbidity and mortality. Sirtuins are anti-aging enzymes that play a diverse role in cellular energy metabolism and gene regulation. Mice deficient in SIRT1 are more susceptible to developing AKI and sirtuin activation is a potential treatment for AKI.

This is a randomized, double-blind, placebo-controlled, stepwise study of escalating doses of Basis (NR/pterostilbene) in patients with AKI. The study will potentially comprise up to four Steps. The purpose of the stepwise approach is to identify the dose of Basis that achieves at least a 50% and up to 100% increase in white blood cell (WBC) content of nicotinamide adenine dinucleotide (NAD+) without side-effects.

During each Step, Basis (5 patients) or placebo (1 patient) will be given twice a day for 2 days. Patients will have frequent blood sampling performed for a 24 hour period following dosing on Day 1 and then at 48 hr. The measurements in blood will include NR/pterostilbene blood concentrations and NAD+ and NAAD (nicotinic acid adenine dinucleotide) concentrations in WBCs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female hospitalized patients, age ≥ 18 years.
2. Patients who have developed AKI (defined by an increase in serum creatinine by ≥0.3 mg/dL within 48 hours; or an increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days).
3. Adequate hematological and liver function, as assessed by the following laboratory requirements:

   1. Hemoglobin ≥10.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1,500/mm3
   3. Platelet count 100,000/mm3
   4. Total bilirubin ≤1.5 x upper limit of normal (ULN).
   5. ALT and AST ≤2.5 x ULN.
4. Able to provide written informed consent in compliance with the Human Investigation Review Committee (IRB).

Exclusion Criteria:

1. Exposure to any investigational agent within 30 days prior to enrollment.
2. Known allergy to any of the study drugs or their excipients.
3. Currently pregnant (confirmed with a positive serum pregnancy test) or nursing.
4. Unstable or clinically significant concurrent medical condition, psychiatric illness or social situation that would, in the opinion of the investigator, jeopardize the safety of a subject and/or their compliance with the protocol.
5. Baseline CKD stage 4-5 (eGFR<30 mL/minute/1.73 m2 as determined using the Modification of Diet in Renal Disease (MDRD) equation; in cases where the MDRD equation may not be suitable, a 24 hour urine creatinine clearance test may be substituted), prior to current hospitalization
6. Any malignancy with the exception of cervical carcinoma in situ,nonmelanoma skin cancer, or superficial bladder tumors that have been successfully and curatively treated with no evidence of recurrent or residual disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration [Cmax] of NR | 2 days
  Maximum plasma concentration [Cmax] of NR after oral administration of Basis
Maximum plasma concentration [Cmax] of pterostilbene | 2 days
  Maximum plasma concentration [Cmax] of pterostilbene after oral administration of Basis
Area Under the Curve [AUC] of NR | 2 days
  Area Under the Curve [AUC] of NR after oral administration of Basis
Area Under the Curve [AUC] of pterostilbene | 2 days
  Area Under the Curve [AUC] of pterostilbene after oral administration of Basis
Incidence of Treatment-Emergent Adverse Events (Safety) | 2 days
  Subjects will be interviewed to determine onset of nausea, abdominal pain, vomiting, diarrhea, or rash. Adverse events will be characterized as probably related, probably not related, or unknown
Incidence of Treatment-Emergent Laboratory Abnormalities (Safety) | 2 days
  comprehensive metabolic panel (including liver function tests), complete blood count

SECONDARY OUTCOMES:
NAD+ levels | 2 days
  To determine the increase in NAD+ levels in white blood cells (WBCs) following twice daily Basis administration
Dose finding for 50% increase in NAD+ levels in WBCs | 2 days
  Dose of Basis that leads to 50% increase in NAD+ levels in WBC
Dose finding for 100% increase in NAD+ levels in WBCs | 2 days
  Dose of Basis that leads to 100% increase in NAD+ levels in WBC

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Rhee, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simic P, Vela Parada XF, Parikh SM, Dellinger R, Guarente LP, Rhee EP. Nicotinamide riboside with pterostilbene (NRPT) increases NAD+ in patients with acute kidney injury (AKI): a randomized, double-blind, placebo-controlled, stepwise safety study of escalating doses of NRPT in patients with AKI. BMC Nephrol. 2020 Aug 13;21(1):342. doi: 10.1186/s12882-020-02006-1. PMID 32791973